CLINICAL TRIAL: NCT04646525
Title: The Relationship Between Mild Covid-19 Infection in Pediatric Patients and Protection of Secondary Lymphoid Organs
Brief Title: The Relationship Between Covid-19 Infection in Pediatric Patients and Secondary Lymphoid Organs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Merih Onal, Assistant Professor, Selcuk University
Other Study IDs: 2020/480
Record Dates: First submitted 2020-11-05; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Covid19; Immune Deficiency; Tonsillitis; Tonsil Hypertrophy; Adenoiditis; Adenoid Hypertrophy
Keywords: pediatric; covid19; İmmune system
MeSH Terms: conditions — COVID-19; Immunologic Deficiency Syndromes; Tonsillitis | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Physical examination — Pediatric patients diagnosed with COVID-19 and who have had infection will be examined, adenoid and tonsillar tissues will be evaluated in terms of hypertrophy, chronic, or recurrent infection.
  Other Names: Only the tonsil and adenoid tissues of the patients will be examined by physical examination, no intervention will be done

SUMMARY:
We aimed to find out whether the tonsils and nasal tissues of pediatric patients are the main factors that protects the children's immune system against COVID-19 infection.

DETAILED DESCRIPTION:
Since it is known that the tonsil and adenoid tissues that are known as a secondary lymphoid organ, which form the first line of defense, are more active in childhood than adults, especially in the childhood age group, and since it has been scientifically shown that patients diagnosed with COVID-19 infection in the pediatric age group overcome this disease lightly than adults, we aimed to reveal whether the defined tonsil and adenoid tissues are the main factors that protect the children's immune system against COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COVID-19 infection.
* Patients aged between 1-16 years
* Patients whose PCR test becomes negative

Exclusion Criteria:

* Patients with lymphoid tissue malignant disease
* Patients with known lung disease
* Patients with known systemic disease

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients between the ages of 1-16 diagnosed with Covid-19 will be examined by the ENT doctor in terms of tonsil and adenoid tissues after they overcome the active infection period and PCR tests turn negative.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of our study was the evaluation of pediatric patients diagnosed with COVID-19 and who had COVID-19 infection in terms of adenoid and tonsillar tissue hypertrophy and the presence of chronic or recurrent infection. | 2020-2021
  The structure of the tonsil and adenoid tissues will be examined by physical examination, and the presence of tonsil and adenoid hypertrophy, tonsillitis, and adenoiditis conditions will be identified. The severity of covid-19 will be determined according to the cases of patients with tonsil and adenoid tissue disorders, who are hospitalized in intensive care, have infiltration in the lungs, and receive oxygen support.

CONTACTS AND LOCATIONS:
Overall Officials: Merih Onal, Assist. Prof., Principal Investigator — Selcuk University
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share our study data after completing collecting patient data and preparing the article about the study.

REFERENCES:
- [Background] Brodin P. Why is COVID-19 so mild in children? Acta Paediatr. 2020 Jun;109(6):1082-1083. doi: 10.1111/apa.15271. Epub 2020 Apr 15. No abstract available. PMID 32212348
- [Background] Dong Y, Mo X, Hu Y, Qi X, Jiang F, Jiang Z, Tong S. Epidemiology of COVID-19 Among Children in China. Pediatrics. 2020 Jun;145(6):e20200702. doi: 10.1542/peds.2020-0702. Epub 2020 Mar 16. PMID 32179660